CLINICAL TRIAL: NCT00308230
Title: A Pilot Study of B-Type Natriuretic Peptide (BNP) Levels in Patients With Congenital Heart Disease and Systemic Right Ventricles or Volume Overloaded Pulmonic Right Ventricles
Brief Title: Pilot Study of B-Type Natrieutic Peptide (BNP) Levels in Patients With Congenital Heart Disease(BNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Wendy M. Book, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00045884
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Congenital Heart Disease; Cardiovascular Disease
Keywords: Congenital, BNP
MeSH Terms: conditions — Heart Defects, Congenital; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Heart (Placebo Comparator): Control Group with Normal Heart
  Interventions: Procedure: Six minute walk test; Behavioral: Minnesota Living with Heart Failure Questionnaire
- Congenital Heart Disease (Active Comparator): Tetralogy of Fallot, DTGA, CCTGA
  Interventions: Procedure: Six minute walk test; Behavioral: Minnesota Living with Heart Failure Questionnaire
- Heart Failure (Active Comparator): Left ventricular heart failure, no congestive heart disease
  Interventions: Procedure: Six minute walk test; Behavioral: Minnesota Living with Heart Failure Questionnaire

INTERVENTIONS:
Procedure: Six minute walk test
Behavioral: Minnesota Living with Heart Failure Questionnaire

SUMMARY:
The object of this study is to measure the levels of B-type Natriuretic Peptide (BNP) in patients with congenital heart disease, normal individuals, and patients with acquired heart failure, and compare the results from each group.

DETAILED DESCRIPTION:
Enrollment: Patients with congenital heart disease seen at Emory Clinics, Adult Congenital Heart Disease program, Crawford Long Hospital will be asked to participate in this pilot study. Sample size: 20 patients (5 in each group) Screening Phase: Demographic data, medical history, physical examination including vital signs and room air oxygen saturation, and medications will be recorded. New York Heart association functional class will be recorded.

BNP Levels: Approximately 7 cc of blood will be collected. The blood will be analyzed for B-type natriuretic peptide on a rapid assay in the clinic.

Exercise Tolerance: will be measured by a 6 minute walk test on day of visit Echocardiogram: A complete echocardiogram including assessment of anatomy, ventricular function and valvular function will be performed following the phlebotomy.

Quality of life: The minnesota living with heart failure questionnaire will be administered on the day of collection of neurohormonal levels. A research nurse will be available to assist the patient if needed.

ELIGIBILITY:
Inclusion Criteria:Patients with a systemic right ventricle and a subpulmonic left ventricle-including patients with transposition of the great arteries (d-TGA) who have undergone Mustard and Senning repairs (atrial switch procedures) and patients with congenitally corrected TGA (l-TGA) Subpulmonic right ventricle in the absence of pulmonary hypertension (repaired tetralogy of Fallot, congenital pulmonic regurgitation) 4-chambered heart Age > 18 years Participants will have either acquired left ventricular dysfunction (ejection fraction < 35%) or no known cardiac disease For the control group, individuals will have normal cardiac anatomy and normal left ventricular function (determined by echocardiogram) and no known cardiac disease.

Exclusion Criteria:

Single ventricle and or single atria Liver disease with portal hypertension Renal disease requiring dialysis Creatine > 4.0 Significant pulmonary hypertension (systolic PAP >60 mmHg by Echo) Uncontrolled systemic arterial hypertension (systolic > 200 mmHg or diastolic >105 mmHg) Myocardial infarction or acute coronary syndrome within 2 months D-TGA status post atrial switch procedure (Jatene) Intracardiac shunts Inadequate echocardiogram windows Coronary Angioplasty 30 days

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2001-12; Primary Completion 2004-03 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Book, M.D., Principal Investigator — Emory University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical specialty clinic
Pre-assignment Details: No washout or run-in period. Participants were stable Ambulatory outpatients with no changes in their medical regimen for prior to enrollment.
  Exclusions included inability to complete a six minute walk, inability to cooperate with instructions, congenital diagnosis other than the three listed in the CHD group (TOF, DTGA, CCTGA)
Groups:
- Control Group: Structurally normal heart without heart disease.
- Congenital Heart Disease: Tetralogy of Fallot, d-transposition of the great arteries, congenitally corrected transposition of the great arteries
- Heart Failure: Acquired left ventricular heart failure, no history of congenital heart disease
Period: Overall Study
Arm/Group | Control Group | Congenital Heart Disease | Heart Failure
Started | 6 | 8 | 20
Completed | 6 | 8 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Structurally normal heart without heart disease
- Total: Total of all reporting groups
Arm/Group | Control | Congenital Heart Disease | Heart Failure | Total
Number analyzed (Participants) | 6 | 8 | 20 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 20 | 34
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 11
  Male | 2 | 5 | 16 | 23

OUTCOME MEASURES:

1. Primary Outcome: BNP Levels
Description: Levels of B-type naturietic peptide in the blood
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Control Group: Structurally normal hearts
- Congenital Heart Disease: TOF, DTGA, CCTGA-tetralogy of Fallot, the transposition of the great arteries, congenitally corrected transposition
- Heart Failure: Left ventricular failure
Arm/Group | Control Group | Congenital Heart Disease | Heart Failure
Number analyzed (Participants) | 6 | 8 | 20
pg/ml | 16.3 (17.3) | 42.4 (44.8) | 384.3 (452.8)

ADVERSE EVENTS:
Arm/Group | Control Group | Congenital Heart Disease | Heart Failure
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/20
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No